CLINICAL TRIAL: NCT04313634
Title: Targeting Cellular Senescence With Senolytics to Improve Skeletal Health in Older Humans: A Phase 2, Single-Center, 20-week, Open-Label, Randomized Controlled Trial.
Brief Title: Targeting Cellular Senescence With Senolytics to Improve Skeletal Health in Older Humans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sundeep Khosla, M.D. (Other)
Responsible Party: Sponsor-Investigator, Sundeep Khosla, M.D., Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-010546
Record Dates: First submitted 2020-03-17; First posted 2020-03-18 (Actual); Results first posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Healthy
MeSH Terms: interventions — Dasatinib; Quercetin; fisetin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dasatinib plus Quercetin Treatment Goup (Experimental): Subjects will receive Dasatinib (D; 100 mg for two days) plus Quercetin (Q; 1000 mg total daily for three consecutive days taken orally on an intermittent schedule (starting every 28 days) with no-therapy periods in between dosing regimens, repeated every 28 days over 20 weeks, resulting in five total dosing periods throughout the entire intervention
  Interventions: Drug: Dasatinib; Drug: Quercetin
- Fisetin Treatment Group (Experimental): Subjects will receive Fisetin (F; ~20 mg/kg/day for three consecutive days) taken orally on an intermittent schedule (starting every 28 days) with no-therapy periods in between dosing regimens, repeated every 28 days over 20 weeks, resulting in five total dosing periods throughout the entire intervention
  Interventions: Drug: Fisetin
- Untreated Control Group (No Intervention): Subjects will not receive any intervention

INTERVENTIONS:
Drug: Dasatinib — Dasatinib will be supplied as 100 mg tablet white to off-white, biconvex, oval, film- coated
  Other Names: Sprycel
  Arms: Dasatinib plus Quercetin Treatment Goup
Drug: Quercetin — Quercetin will be supplied as quercetin phytosome (sophora japonica concentrate (leaf) / phosphatidylcholine complex from Sunflower) 250 mg
  Arms: Dasatinib plus Quercetin Treatment Goup
Drug: Fisetin — Fisetin will be supplied in 100 mg capsules to be administered orally
  Arms: Fisetin Treatment Group

SUMMARY:
To determine if senolytic drugs reduce senescent cell burden and reduce bone resorption markers/increase bone formation markers in elderly women.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide informed consent.
* Normal postmenopausal women
* Aged ≥60 years

Exclusion Criteria:

* Hemoglobin A1c ≥8.0% at screening
* Subjects who are type II diabetic and on insulin
* Abnormal screening labs: Calcium >10.1 mg/dL, Phosphorus >4.7 mg/dL, Thyroid stimulating hormone (TSH) level <0.3mU/L, Fasting blood glucose >200 mg/dL.
* Presence of significant liver (total bilirubin, AST, ALT, or alkaline phosphatase >2x upper normal limit) or kidney disease (eGFR<30 ml/min/1.73 m2 (using the cystatin C blood levels for analysis). If any elevation were to be noted (2x the normal limit), the study participant would stop treatment and have levels re-drawn in a month, per the clinical judgement of the investigator
* Presence of a clinical diagnosis of heart failure
* Known active malignancy (including myeloma)
* Current diagnosis of malabsorption or undergoing treatment for malabsorption disease
* If any of the laboratory blood work drawn at the study visits return with lab values outside of the "normal limits" or show a significant change from a previous value, a repeat blood draw would be done before the subject is excluded.
* Gastric bypass/reduction
* Hyperthyroidism
* Acromegaly
* Cushing's syndrome
* Hypopituitarism
* Subjects with a fracture within the past six months
* Undergoing treatment with any medications that affect bone turnover, including the following:

  * adrenocorticosteroids (> 3 months at any time or > 10 days within the previous yr, except for use of topical steroid creams or gels or inhaled steroids), anticonvulsant therapy (within the previous year), include only those taking Carbamazepine, Phenobarbital and Phenytoin,
  * bisphosphonates (within the past 3 yrs),
  * denosumab,
  * estrogen (E) therapy or treatment with a selective E receptor modulator, or teriparatide (within the past yr)
* QTc >450 msec
* Inability to provide consent
* Inability to tolerate oral medication
* Current diagnosis of hypo- or hyperparathyroidism or currently undergoing treatment for the disease
* Subjects on therapeutic doses of anti-coagulants (e.g. warfarin, heparin, low molecular weight heparin, factor Xa inhibitors, etc)
* Subjects with hypovitaminosis D (25-hydroxyvitamin D [25(OH)D] <20 ng/ml, whose level does not improve above 20 ng/ml after two courses of 4-week treatment of 50,000 IU/d of Vitamin D. They will be referred to their primary provider should this occur.
* Subjects taking anti-arrhythmic medications known to cause QTc prolongation
* Subjects taking potentially senolytic agents within the last 6 months: Quercetin, Luteolin, Dasatinib, Piperlongumine, or Navitoclax
* Subjects currently taking drugs that induce cellular senescence: alkylating agents, anthracyclines, platins, other chemotherapy
* Subjects taking H2 antagonists, unless randomized to the control group
* Tyrosine kinase inhibitor therapy
* Subjects not having a PBTL p16INK4a mRNA expression level >95 percentile of young female controls (this cut-off is depicted by the dotted line in Fig. 6)
* Known hypersensitivity or allergy to Dasatinib orQuercetin
* Subjects taking the following antimicrobial agents: Aminoglycosides, Azole antifungals (fluconazole, miconazole, voriconazole, itraconazole), Macrolides (clarithromycin, erythromycin), Antivirals (nelfinavir, indinavir, saquinavir, ritonavir, elbasvir/grazoprevir), Rifampin
* If the DXA assessment reveals a spine or femur neck T-score < -2.5, the participant will be advised of this. She would then be given the option of withdrawing from the study to immediately start an osteoporosis drug through her primary care physician or continue in the study and defer osteoporosis drug treatment for the duration of the study (20 weeks). Given that osteoporosis is a chronic, long-term disease, the 20-week deferral would pose a minimal risk to the participant and she would be free to make this choice.
* Subjects taking medications that are sensitive to substrates or substrates with a narrow therapeutic range for CYP3A4, CYP2C8, CYP2C9, or CYP2D6 or strong inhibitors or inducers of CYP3A4 (e.g., cyclosporine, tacrolimus or sirolimus). If antifungals are necessary from an infectious disease perspective, then they will be allowed only if the levels are therapeutic.
* Subjects taking strong inhibitors of CYP3A4
* Subjects on antiplatelet agents (Clopidogrel [Plavix]; Dipyridamole + Asprin [Aggrenox]; Ticagrelor [Brilinta]; Prasugrel [Effient]; Ticlopidine [Ticlid] or Other) who are unable or unwilling to reduce or hold therapy prior to and during the study drug dosing periods. Subjects may continue their previous regimen between study drug dosing periods.
* Subjects on quinolone antibiotic therapy for treatment or for prevention of infections within ten days.
* Subjects taking proton pump inhibitors and unwilling to discontinue therapy for two days before and during the study drug dosing periods.
* Subjects with clinically evident fluid retention
* Subjects with evidence of right heart strain on ECG
* Subjects with a history of pulmonary hypertension
* Subjects with an abnormal Complete Blood Count (clinically insignificant changes would be acceptable based on the judgement of the investigators)
* Presence of any condition the Investigator believes would place the subject at risk or would preclude the subject from successfully completing all aspects of the trial.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sundeep Khosla, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Farr JN, Monroe DG, Atkinson EJ, Froemming MN, Ruan M, LeBrasseur NK, Khosla S. Characterization of Human Senescent Cell Biomarkers for Clinical Trials. Aging Cell. 2025 May;24(5):e14489. doi: 10.1111/acel.14489. Epub 2025 Jan 17. PMID 39823170
- [Derived] Farr JN, Atkinson EJ, Achenbach SJ, Volkman TL, Tweed AJ, Vos SJ, Ruan M, Sfeir J, Drake MT, Saul D, Doolittle ML, Bancos I, Yu K, Tchkonia T, LeBrasseur NK, Kirkland JL, Monroe DG, Khosla S. Effects of intermittent senolytic therapy on bone metabolism in postmenopausal women: a phase 2 randomized controlled trial. Nat Med. 2024 Sep;30(9):2605-2612. doi: 10.1038/s41591-024-03096-2. Epub 2024 Jul 2. PMID 38956196

RESULTS

PARTICIPANT FLOW:
Groups:
- Dasatinib Plus Quercetin Treatment Goup: Subjects received Dasatinib (D; 100 mg for two days) plus Quercetin (Q; 1000 mg total daily) for three consecutive days taken orally on an intermittent schedule (starting every 28 days) with no-therapy periods in between dosing regimens, repeated every 28 days over 20 weeks, resulted in five total dosing periods throughout the entire intervention
  Dasatinib: Dasatinib will be supplied as 100 mg tablet white to off-white, biconvex, oval, film- coated
  Quercetin: Quercetin will be supplied as quercetin phytosome (sophora japonica concentrate (leaf) / phosphatidylcholine complex from Sunflower) 250 mg
- Fisetin Treatment Group: Subjects received Fisetin (F; ~20 mg/kg/day for three consecutive days) taken orally on an intermittent schedule (starting every 28 days) with no-therapy periods in between dosing regimens, repeated every 28 days over 20 weeks, resulted in five total dosing periods throughout the entire intervention
  Fisetin: Fisetin will be supplied in 100 mg capsules to be administered orally
- Untreated Control Group: Subjects did not receive any intervention
Period: Overall Study
Arm/Group | Dasatinib Plus Quercetin Treatment Goup | Fisetin Treatment Group | Untreated Control Group
Started | 30 | 14 | 30
Completed | 27 | 12 | 28
Not Completed | 3 | 2 | 2
Not completed — Adverse Event | 2 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dasatinib Plus Quercetin Treatment Goup | Fisetin Treatment Group | Untreated Control Group | Total
Number analyzed (Participants) | 30 | 14 | 30 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.2 (4.9) | 75.9 (3.7) | 74.4 (6.7) | 73.7 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 14 | 30 | 74
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 30 | 14 | 30 | 74
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 29 | 14 | 30 | 73
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 14 | 30 | 74

OUTCOME MEASURES:

1. Primary Outcome: Change in C-terminal Telopeptide of Type I Collagen [CTX]
Description: Percent change in serum bone turnover markers C-terminal telopeptide of type I collagen [CTX]. The C-terminal telopeptide (CTX), also known as carboxy-terminal collagen crosslinks, is a biomarker used to measure the rate of bone turnover. It provides valuable information for assessing bone health and evaluating treatment responses.
Time Frame: Baseline, 20 weeks
Measure: Median (Full Range); unit: percent change
Arm/Group | Dasatinib Plus Quercetin Treatment Goup | Fisetin Treatment Group | Untreated Control Group
Number analyzed (Participants) | 28 | 11 | 28
percent change | -4.1 [-28.1 to 114.6] | 13.7 [-42.7 to 61.0] | -7.7 [-42.4 to 22.5]
Statistical Analysis 1: Comparison: Dasatinib Plus Quercetin Treatment Goup vs Untreated Control Group; Test type: Superiority; p = 0.611, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in Bone Turnover Markers
Description: Percent change in amino-terminal propeptide of type I collagen (P1NP). The P1NP assay measures the serum concentration of the amino-terminal propeptide of type I procollagen (P1NP). As the concentration of this extension propeptide is directly proportional to the amount of new collagen laid down in bone, it can be used to assess bone formation.
Time Frame: Baseline, 2 weeks
Measure: Median (Full Range); unit: percentage change of P1NP
Arm/Group | Dasatinib Plus Quercetin Treatment Goup | Fisetin Treatment Group | Untreated Control Group
Number analyzed (Participants) | 30 | 11 | 30
percentage change of P1NP | 0.8 [-39.6 to 113.5] | -31.9 [-74.0 to 23.3] | -15.2 [-55.0 to 59.8]
Statistical Analysis 1: Comparison: Dasatinib Plus Quercetin Treatment Goup vs Untreated Control Group; Test type: Superiority; p = 0.020, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Bone Turnover Markers
Description: as for outcome 2
Time Frame: Baseline, 4 weeks
Population: Outcome measure was only collected and reported for Dasatinib plus Quercetin Treatment arm and Untreated Control group arm
Measure: Median (Full Range); unit: percentage change of P1NP
Arm/Group | Dasatinib Plus Quercetin Treatment Goup | Untreated Control Group
Number analyzed (Participants) | 29 | 30
percentage change of P1NP | 4.2 [-61.4 to 1480] | -12.1 [-58.0 to 95.9]
Statistical Analysis 1: Comparison: Dasatinib Plus Quercetin Treatment Goup vs Untreated Control Group; Test type: Superiority; p = 0.024, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Bone Turnover Markers
Description: as for outcome 2
Time Frame: Baseline, 20 weeks
Measure: Median (Full Range); unit: percentage change of P1NP
Arm/Group | Dasatinib Plus Quercetin Treatment Goup | Fisetin Treatment Group | Untreated Control Group
Number analyzed (Participants) | 28 | 11 | 28
percentage change of P1NP | -8.6 [-48.1 to 130.9] | 4.5 [-34.8 to 29.7] | 0.1 [-49.2 to 95.2]
Statistical Analysis 1: Comparison: Dasatinib Plus Quercetin Treatment Goup vs Untreated Control Group; Test type: Superiority; p = 0.149, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in Bone Mineral Density (BMD)
Description: Percent change in BMD by dual-energy X-ray absorptiometry (DXA) at the lumbar spine, hip ((total and femoral neck (FN), and radius (total and ultra-distal)).
Time Frame: Baseline, 20 weeks
Population: Each skeletal site was measured and assessed separately. As such, some sites (which are influenced by osteoarthritis) did not provide interpretable scans. This occurred due to motion artifacts or other issues. Therefore, the number of participants analyzed differ by skeletal site.
Measure: Median (Full Range); unit: percentage of change in BMD
Arm/Group | Dasatinib Plus Quercetin Treatment Goup | Fisetin Treatment Group | Untreated Control Group
Number analyzed (Participants) | 28 | 12 | 29
percentage of change in BMD
  Lumbar Spine: number analyzed (Participants) | 22 | 11 | 24
  Lumbar Spine | -0.2 [-3.1 to 6.2] | 0 [-1.5 to 8.9] | 0.5 [-10.4 to 6.8]
  Hip (Femoral neck ) | -0.3 [-4.8 to 4.0] | -0.9 [-3.7 to 2.0] | -0.5 [-6.0 to 19.2]
  Radius: number analyzed (Participants) | 27 | 12 | 28
  Radius | 0.4 [-3.0 to 6.9] | 0.7 [-12.1 to 5.7] | 0.2 [-4.7 to 12.9]

6. Secondary Outcome: Change in Plasma Senescence-associated Secretory Phenotype (SASP)
Description: Percent change in SASP cells (representing the total senescence cell burden) present. Assessment of senescence markers in bone at baseline and 2 weeks.
Time Frame: Baseline, 2 weeks
Measure: Median (Full Range); unit: percent change
Arm/Group | Dasatinib Plus Quercetin Treatment Goup | Fisetin Treatment Group | Untreated Control Group
Number analyzed (Participants) | 30 | 11 | 30
percent change | -2.6 [-187.7 to 16.4] | -0.9 [-41.8 to 3.7] | -2.5 [-110.4 to 91.5]
Statistical Analysis 1: Comparison: Dasatinib Plus Quercetin Treatment Goup vs Untreated Control Group; Test type: Superiority; p = 0.953, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study, approximately 20 weeks
Arm/Group | Dasatinib Plus Quercetin Treatment Goup | Fisetin Treatment Group | Untreated Control Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/14 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 1/14 | 0/30
Other Adverse Events (participants affected / at risk) | 23/30 | 12/14 | 5/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib Plus Quercetin Treatment Goup (N=30) | Fisetin Treatment Group (N=14) | Untreated Control Group (N=30)
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib Plus Quercetin Treatment Goup (N=30) | Fisetin Treatment Group (N=14) | Untreated Control Group (N=30)
Abdominal distention (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 7 (14) | 1 (1) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nausea (General disorders) | 5 (8) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Covid (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Metabolism and nutrition disorders - other (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac disorders - other (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 16 (36) | 1 (1) | 0 (0)
Muscle weakness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - other (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Facial pain (General disorders) | 1 (4) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (8) | 1 (2) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 3 (4) | 1 (2) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 1 (2) | 0 (0)
Hot flashes (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders - other (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (4) | 1 (1) | 1 (1)
Cataract surgery (Eye disorders) | 1 (2) | 1 (2) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (10) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-08): https://cdn.clinicaltrials.gov/large-docs/34/NCT04313634/Prot_SAP_000.pdf